CLINICAL TRIAL: NCT02215655
Title: Increasing Autonomous Motivation in ESRD to Enhance Phosphate Binder Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Ebele Umeukeje, Fellow, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 141143
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease
Keywords: phosphate binder adherence; autonomous motivation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing (Active Comparator): Motivational interviewing counselling will be administered to the subjects
  Interventions: Behavioral: Motivational interviewing
- No intervention: control group (No Intervention): No motivational interviewing counselling will be administered to the subjects

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing counselling sessions will be administered to the subjects.
  Arms: Motivational interviewing

SUMMARY:
Hyperphosphatemia in end-stage renal disease (ESRD) patients is a non-traditional risk factor for all-cause and cardiovascular mortality. Non-adherence to phosphate binders is as high as 74% in ESRD patients and has been shown to be most related to psychosocial factors including attitudes. There is limited data on the influence of attitudes and perceived autonomy support on phosphate binder adherence and these two psychosocial constructs can be positively influenced through the use of motivational interviewing skills to increase autonomous motivation. Furthermore, racial disparities are known to exist in ESRD however and there are still gaps, which exist in understanding the determinants of disparities in adherence in vulnerable patients with ESRD.

In this study, the investigators seek to determine the impact of motivational interviewing on phosphate binder adherence in diverse ESRD patients. The investigators will ask all the subjects to fill out surveys mainly regarding their attitudes; perceived providers' autonomy support and phosphate binder adherence. The investigators will administer motivational counseling to subjects in the intervention arm of the study, at baseline and 1 month after recruitment. The investigators will ask all the subjects to fill out the same surveys 2 months after recruitment and the investigators will compare subjects who underwent motivational interviewing to those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Receiving phosphate binder therapy currently
* English speaking

Exclusion Criteria:

* Non- English speaking
* Known diagnosis of psychosis or dementia, limiting ability to provide informed consent
* Any medical condition that precludes participation in the study including deafness, dying etc.
* Initial Morisky Medication Adherence score greater than 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
change in subjects' adherence to phosphate binders | baseline and 2 months
  Change from baseline in the following survey at 2 months:
  - Morisky Medication Adherence Scale (MMAS)

SECONDARY OUTCOMES:
change in attitudes towards phosphate binder therapy | baseline and 2 months
  Change from baseline in the following survey/questionnaire at 2 months:
  - Autonomous Regulation Scale (AR)
change in perceived providers' autonomy support towards phosphate binder therapy | baseline and 2 months
  Change from baseline in the following survey/questionnaire at 2 months:
  - Health Care Climate Questionnaire (HCC)

CONTACTS AND LOCATIONS:
Overall Officials: Ebele M Umeukeje, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States